CLINICAL TRIAL: NCT04468542
Title: Randomized Placebo-controlled Analysis of Superior Laryngeal Nerve Block for Neurogenic Cough
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Anthony Grady, Principal investigator (physician), University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY001182
Record Dates: First submitted 2020-07-07; First posted 2020-07-13 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Cough; Nerve Block
Keywords: Superior laryngeal nerve; Neurogenic cough; Nerve Block; Idiopathic cough
MeSH Terms: conditions — Cough | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bupivacaine/triamcinolone injection (Experimental): 2-cc injection (mixture consisting of 1-cc of 0.5% Bupivacaine injection and 1cc of 40mg/cc triamcinolone acetonide suspension injection) will be delivered percutaneously into the region of the proximal superior laryngeal nerve, every 1-2 weeks, for total of 2 to 3 injections
  Interventions: Drug: Superior laryngeal nerve block - Intervention (Bupivacaine and triamcinolone acetonide suspension)
- Saline injection (Placebo Comparator): 2-cc injection of normal saline will be delivered percutaneously into the region of the proximal superior laryngeal nerve, every 1-2 weeks, for total of 2 to 3 injections
  Interventions: Drug: Superior laryngeal nerve block - Placebo (saline)

INTERVENTIONS:
Drug: Superior laryngeal nerve block - Intervention (Bupivacaine and triamcinolone acetonide suspension) — 2-cc injection (mixture consisting of 1-cc of 0.5% Bupivacaine injection and 1cc of 40mg/cc triamcinolone acetonide suspension injection) will be delivered percutaneously into the region of the proximal superior laryngeal nerve, every 1-2 weeks, for total of 2 to 3 injections
  Arms: Bupivacaine/triamcinolone injection
Drug: Superior laryngeal nerve block - Placebo (saline) — 2-cc injection of saline will be delivered percutaneously into the region of the proximal superior laryngeal nerve, every 1-2 weeks, for total of 2 to 3 injections
  Arms: Saline injection

SUMMARY:
Prospective randomized placebo-controlled trial assessing the efficacy of superior laryngeal nerve block for adults with neurogenic cough refractory to proton pump inhibitor as determined by improvement in validated cough severity questionnaires before and after injection of Marcaine and Kenalog compared to placebo (saline injection).

DETAILED DESCRIPTION:
Abbreviations/ Definitions: cough severity index (CSI), Cough quality of life questionnaire (CQLQ), proton pump inhibitor (PPI), nasopharyngolaryngoscopy (NPL), University of South Florida (USF), superior laryngeal nerve (SLN), upper airway cough syndrome (UACS), food and drug administration (FDA), investigational new drug (IND), medical record number (MRN), electronic medical record (EMR), ear nose and throat (ENT), angiotensin converting enzyme (ACE), chronic rhinosinusitis (CRS), gastroesophageal reflux disorder (GERD), pulmonary function test (PFT), Reflux finding score (RFS), Speech and language pathology (SLP)

Participants will be referred into (via other USF affiliated departments) or recruited within the University of South Florida Department of Otolaryngology practice. Individuals will be screened for eligibility based on referral description. Eligibility will be determined by history at initial visit based on inclusion and exclusion criteria. Eligible participants will be adults with chronic cough >8 weeks duration and presumed neurogenic cough based on initial evaluation. Chronic throat clearing with foreign body sensation for >8 weeks duration will also meet criteria for inclusion and will be used synonymously with and considered chronic cough for the remainder of this protocol and study. Patients will be excluded if primary cause is determined to not be neurogenic. Patients will be excluded if there are other possible significant contributors to the cough that have not been treated (no other obvious treatable and untreated cause), or they will be treated per the standard of care prior to enrolling in this study. Patients will be screened for at least a 4-week course of PPI therapy during duration of symptoms. Patients with possible UACS were included if a trial of medications had been completed previously. If patients are on long term medications that are effective for their respective related condition (but still ineffective at adequately controlling chronic cough), they will be encouraged to make no unnecessary changes through treatment/study duration. These include acid suppression therapy (outside of the recent 6-week trial of PPI if applicable), therapy for UACS symptoms if indicated (eg, Flonase and antihistamine, saline rinses, etc.), neuromodulators (e.g., gabapentin). Patients were excluded if they started any of these medications in last month and were not willing to discontinue them for the duration of the trial. Participants must be willing and able to consent to participate in the study, be willing to be assigned to and undergo intervention or the placebo, and be willing to adhere to the study protocol for the duration of the trial: 2-4 visits, approximately 3 weeks of treatment, 6 week PPI trial with 4 week discontinuation period if no improvement (if applicable), up to 12 week follow up questionnaires (survey only), participate in cough suppression, take PPI as prescribed for duration specified.

Participants were excluded if at any point they met the following criteria: unwilling to participate in protocol, allergic to Bupivacaine or triamcinolone acetonide suspension, presence of severe uncontrolled medical condition, any significant pulmonary processes (including chronic obstructive pulmonary disease, bronchiectasis, non-asthmatic eosinophilic bronchitis, structural abnormalities, etc.), presence of asthma (determined by presence of abnormal pulmonary function test (PFT) provocation testing), concern for aerodigestive tract malignancy from history or exam, structural abnormality seen on NPL or prior imaging, immunocompromised, current smoker, use of ACE inhibitor at time of or one month preceding first injection, or vulnerable population.

Eligible participants underwent NPL will be also conducted at initial visit (Reflux finding score, RFS). Informed consent will be obtained at this time. Demographics (including sex, age, past medical history, related comorbidities, sidedness of globus sensation, neuromodulator use, results of any prior chest radiograph during symptom duration, ever referred to SLP for voice therapy) will be recorded at initial visit. Related comorbidities include UACS, allergic rhinitis, CRS, GERD. Patients who had not previously received adequate PPI trial were placed in 4 to 6-week course and encourage/counseled to complete lifestyle modifications to reduce reflux. Patients with less than complete response to PPI (persistent clinically significant cough) therapy were included in study. Patients follow-up visit for consideration of injection was schedule one month after discontinuing PPI trial. Questionnaire scores were determined immediately prior to first injection. All patients were counseled on cough suppression prior to initial injection. Patients were randomly assigned to placebo (2-cc normal saline) or intervention (total of 2-cc injection, mixture consisting of 1-cc of Bupivacaine and 1-cc of Kenolog-40) injection groups using computer-generated random assignment. Injections will begin at initial visit or at follow-up visit if trial of PPI required. Immediately preceding injections, patients will be given 5 sprays of 4% topical lidocaine to facilitate injection which will also act to facilitate patient blinding. Injection will be delivered into the region of the proximal superior laryngeal nerve using greater cornu of hyoid and superior cornu of thyroid cartilage as landmarks. Injection will be placed 1-cm anterior to the midpoint of these landmarks.

If globus sensation or trigger site was localized to one side, this was recorded and initial injection was directed at this side, otherwise this was picked at random. The second injection was directed at the same side if partial improvement (patient's subjective sense of least 50% reduction of symptoms) was observed after the first injection. The second injection was directed at the contralateral side if there was no initial improvement. Third injection was offered if there was improvement during either of the first two injections (completed on the ipsilateral side of prior two injections or the side with most improvement if bilateral had been completed). There was no second/third injection if complete resolution of symptoms was observed after the preceding injection. Follow up for repeat injection will be scheduled in 1-2 weeks, and exact time recorded. Questionnaire scores were then recorded 2 weeks after final injection of the series. Surveys (see next section, CSI and CQLQ) will also be sent for patients to complete at 6 and 12 weeks after last injection, which will be analyzed in subsequent study. Surveys will have a one-week window to be considered in their nominal category. All adverse events will be recorded. See data capture sheet for collected variables.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults referred into or treated by the University of South Florida department of Otolaryngology practice with chronic cough (including throat clearing with globus) as determined by presence > 8 weeks duration
* Presumed to have neurogenic component based on history with no other obvious treatable (and untreated) cause
* refractory to proton pump inhibitor (PPI) therapy (at least 4 week trial)
* no improvement of upper airway cough syndrome symptoms with medications if indicated (eg, Flonase and antihistamine)
* Patients may continue any medications for possibly related conditions (e.g., Flonase, gabapentin, etc.) including allergies, chronic sinusitis, acid reflux; there should be NO changes to mediation regimen within 1 months of study initiation (with the exception of patients who were not previously on PPI that failed trail of PPI which they will discontinue 1 month prior to first intervention)
* Willingness to participant be assigned and adhere to the protocol. Participants must be willing and able to consent to participate in the study, be willing to undergo intervention or the placebo, and be willing to commit to adhere to the study protocol for the duration of the trial (PPI trial if applicable, 2-4 visits, follow up questionnaires, participate in cough suppression)

Exclusion Criteria:

* unwilling to participate in protocol
* allergic to Marcaine/lidocaine or predisposing condition to allergy
* uncontrolled medical condition (this will be treated on a case by case basis using clinical judgment of risks and the medical condition, with participants being excluded who have conditions that may significantly increase the odds of having a serious or life-threatening reaction)
* pulmonary processes (including chronic obstructive pulmonary disease (chronic obstructive pulmonary disease), bronchiectasis, non-asthmatic eosinophilic bronchitis, structural abnormalities, etc.)
* asthma (must have history of abnormal pulmonary function provocation testing)
* structural abnormality laryngoscopy (this does not pertain to inflammatory findings)
* immunocompromised
* current smoker (>1 cigarette in past month)
* use of angiotensin converting enzyme inhibitor current or within past month
* Vulnerable population: students, employees, socially or economically disadvantaged, wards of the state, pregnant women, cognitively impaired adults, non-adults.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
2 week post-treatment cough severity index score improvement | Immediately pre-treatment and post-treatment at 2 weeks
  Measure of efficacy of intervention by comparing change in pre-treatment and 2 week post-treatment cough severity index scores between intervention to placebo
2 week post-treatment cough-specific quality-of-life questionnaire score improvement | Immediately pre-treatment and post-treatment at 2 weeks
  Measure of efficacy of intervention by comparing change in pre-treatment and 2 week post-treatment cough-specific quality-of-life questionnaire scores between intervention to placebo

SECONDARY OUTCOMES:
6 week post-treatment cough severity index score improvement | Immediately pre-treatment and post-treatment at 6 weeks
  Measure of efficacy of intervention by comparing change in pre-treatment and 6 week post-treatment cough severity index scores between intervention to placebo
12 week post-treatment cough severity index score improvement | Immediately pre-treatment and post-treatment at 12 weeks
  Measure of efficacy of intervention by comparing change in pre-treatment and 12 week post-treatment cough severity index scores between intervention to placebo
6 week post-treatment cough-specific quality-of-life questionnaire score improvement | Immediately pre-treatment and post-treatment at 6 weeks
  Measure of efficacy of intervention by comparing change in pre-treatment and 6 week post-treatment cough-specific quality-of-life questionnaire scores between intervention to placebo
12 week post-treatment cough-specific quality-of-life questionnaire score improvement | Immediately pre-treatment and post-treatment at 12 weeks
  Measure of efficacy of intervention by comparing change in pre-treatment and 12 week post-treatment cough-specific quality-of-life questionnaire scores between intervention to placebo

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida South Tampa Clinic, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simpson CB, Tibbetts KM, Loochtan MJ, Dominguez LM. Treatment of chronic neurogenic cough with in-office superior laryngeal nerve block. Laryngoscope. 2018 Aug;128(8):1898-1903. doi: 10.1002/lary.27201. Epub 2018 Apr 18. PMID 29668037
- [Background] Dhillon VK. Superior laryngeal nerve block for neurogenic cough: A case series. Laryngoscope Investig Otolaryngol. 2019 Jul 5;4(4):410-413. doi: 10.1002/lio2.292. eCollection 2019 Aug. PMID 31453350